CLINICAL TRIAL: NCT05935995
Title: Intraoperative Assessment of Surgical Margins Using Confocal Microscopy in Comparison With Reference Extemporaneous Examination (Pilot Study)
Brief Title: Intraoperative Assessment of Surgical Margins Using Confocal Microscopy in Comparison With Reference Extemporaneous Examination
Acronym: HISTOBLOC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-A00818-37
Record Dates: First submitted 2023-06-27; First posted 2023-07-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Basal Cell Carcinoma of Skin
Keywords: margin surgical; confocal microscopy; conventional histopathology (H&E)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Basal Cell; Margins of Excision | interventions — Microscopy, Confocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microscopy confocal (Experimental)
  Interventions: Other: microscopy confocal (Histolog Scanner)

INTERVENTIONS:
Other: microscopy confocal (Histolog Scanner) — Surgical margins of tumor samples will be examined by conventional histopathology (H&E) and confocal microscopy (Histolog® scanner, SamanTree Medical, Switzerland).
  Depending on the histopathological result obtained between the two methods, the patient may benefit directly from early surgery if the experimental result confirms the presence of positive margins (excluding the learning curve).
  A learning curve will be established over the first fifteen surgeries, enabling surgical teams to gain experience and systematize specimen flattening. This learning curve will also enable reference images to be produced. The procedure will be carried out by the surgeon and the pathologist in the operating room during this phase.

SUMMARY:
Study to evaluate the use of confocal microscopy for detecting resection margins in patients undergoing surgery for basal cell carcinoma of skin and squamous Cell Carcinoma of Head and Neck

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥18 years old
* Squamous cell or basal cell tumor (1 to 4 cm) of mucous or cutaneous origin.
* Patient whose surgical indication has been validated in a consultation meeting
* Patients with scheduled surgery
* WHO< or =2
* ASA < 3
* Patient affiliated to the social security system
* Patient has understood, signed and dated the consent form.

Exclusion Criteria:

* History of irradiation in the surgical area
* Women who are pregnant or who are breast-feeding.
* Persons deprived of their liberty or under guardianship (including curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-06-21 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Confocal Microscopy Diagnosis Compared to Gold Standard | 1 day
  The concordance of intraoperative diagnosis between the two methods will be assessed by the condition of the margins of surgical specimens. Diagnostic accuracy will be measured by the sensitivity and specificity of confocal microscopy, using conventional histology reports from extemporaneous examination as the gold standard.
  * negative margins (absence of tumour cells) ;
  * positive margins (presence of tumour cells).

CONTACTS AND LOCATIONS:
Overall Officials: GILLES DOLIVET, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No